CLINICAL TRIAL: NCT05252663
Title: Effect of Intrathorathic Oscillations on Pulmonary Functions in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Elsayed Abbass, Dr.Mai Elsayed Abbass, Lecturer of pediatric physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/012/003589
Record Dates: First submitted 2022-02-13; First posted 2022-02-23 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Quake breathing, patients were advised to take a deep breath and hold it for 3-5 seconds.
  Interventions: Procedure: Quake device training
- Control group (Active Comparator): Percussion, vibration and shaking were used accompanied with postural drainage.
  Interventions: Procedure: Traditional chest physiotherapy

INTERVENTIONS:
Procedure: Quake device training — In Quake breathing, patients were advised to take a deep breath and hold it for 3-5 seconds. The patient had the mouthpiece firmly sealed to the lips and were asked to inhale and exhale completely
  Arms: Study group
Procedure: Traditional chest physiotherapy — postural drainage - percussion
  Arms: Control group

SUMMARY:
Aim: To investigate the effect of intrathoracic oscillations on forced expiratory volume at first second and peak expiratory flow in the children with cerebral palsy.

Methods and Procedures: Children were randomly assigned into two groups (study group and control group). Each child was evaluated before and after 6 successive weeks.

DETAILED DESCRIPTION:
Methods and Procedures: 24 children with spastic cerebral palsy from both sexes, There ages from 6 to 8 years old. Children were randomly assigned into two groups (study group and control group). Each child was evaluated before and after 6 successive weeks. The children of the control group received traditional chest physiotherapy. while, the children of the study group received 4 sessions per week for 6 weeks with quake device.

ELIGIBILITY:
Inclusion Criteria:

* children with cerebral palsy
* Age from 6 to 8 years old
* the degree of spasticity from 2 to 2+
* grade 4, 5 according to GMFCs

Exclusion Criteria:

* Uncontrolled convulsions
* Any psychiatric disorders

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2022-06-26 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
FEV1 | After 6 weeks
  Forced expiratory volume at first second
PEF | After 6 weeks
  Peak expiratory flow

CONTACTS AND LOCATIONS:
Overall Officials: Mai Abbass, Ph.D., Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Faculty of Physical Therapy, Cairo University, Cairo
  - Faculty of physical therapy, Cairo university, Cairo

IPD SHARING:
Plan to Share IPD: No